CLINICAL TRIAL: NCT03296488
Title: A Randomized Controlled Trial to Compare the Efficacy and Safety of NALDEBAIN With Intravenous Patient-Controlled Analgesia With Fentanyl for the Treatment of Post-Laparotomy Surgery
Brief Title: The Efficacy and Safety of NALDEBAIN for the Treatment of Post-Laparotomy Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20170089
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Pain, Postoperative
Keywords: post-laparotomy wound pain; NALDEBAIN (150 mg Nalbuphine Sebacate); PCA (patient-control-ed alagesia)
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nalbuphine Sebacate (Experimental): receive single dose of NALDEBAIN (150 mg Nalbuphine Sebacate, 75 mg/ml, 2 ml/vial) intramuscularly 24±12 hours before surgery.
  Interventions: Drug: Nalbuphine Sebacate
- Fentanyl Citrate (Active Comparator): receive intravenous patient-controlled analgesia with fentanyl through 48 hours after surgery.
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Nalbuphine Sebacate — intramuscular single dose of NALDEBAIN 24±12 hours before surgery.
  Other Names: NALDEBAIN
  Arms: Nalbuphine Sebacate
Drug: Fentanyl Citrate — Intravenous patient-controlled analgesia with fentanyl through 48 hours after surgery.
  Other Names: PCA with fentanyl
  Arms: Fentanyl Citrate

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of single doses of intramuscular NALDEBAIN on patients scheduled to undergo elective laparotomy. This will be performed by administering NALDEBAIN pre-operatively to subjects scheduled to undergo elective laparotomy, and assessing the safety and efficacy of the drug compared to PCA with fentanyl. The study will demonstrate whether single use of NALDEBAIN is noninferior to PCA with fentanyl or not.

DETAILED DESCRIPTION:
Screening (Days -30 to -1) (All Study Subjects)

The nature of the study, as well as the potential risks and benefits associated with study participation, will be fully explained to all potential subjects. The following will then be obtained:

* Informed consent.
* Demographic information, including sex, age, BMI and type of surgery.
* Vital signs, including temperature, respiratory rate, blood pressure and heart rate.
* Medical history, including medication use and history of allergy.
* Physical examination.
* Laboratory testing, including hematological and biochemical tests, and urinalysis.
* ECG and X-ray.

Study Day -1 (All Eligible Subjects)

* Eligible subjects will be required to check into the clinical site before surgery (Day -1). The following procedures will be performed upon check-in:

  * Review inclusion/exclusion criteria
  * Randomization
  * Review of concomitant medications
  * Review of adverse events
* Additional laboratory tests will be requested as needed deciding by the investigator.
* All eligible subjects will hospitalize and be randomized into one of two treatment groups:

  * Group 1 - Intramuscular NALDEBAIN.
  * Group 2 - Intravenous PCA with fentanyl. Group 1 will receive single dose of NALDEBAIN (150 mg Nalbuphine Sebacate) intramuscularly 24±12 hours before surgery.

Group 2 will receive intravenous patient-controlled analgesia with fentanyl through 48 hours after surgery.

* Pain assessment: group 1 and 2 will rate their pain intensity using a VAS pain scale prior dosing or at Day -1 respectively.
* Brief Pain Inventory (BPI) will be evaluated at Day -1.
* Vital signs will be checked prior to dosing and once daily before Day 6.
* Group 1 received NALDEBAIN will evaluate injection site within 1 hour prior to dosing.

Study Day 0-5 All subjects will be given general anesthesia prior to their scheduled surgical procedure.

If patients need additional medication for treatment of pain, Ketorolac and Morphine could be used as supplemental analgesics when they needed.

After surgery, the following evaluations will be performed:

* Pain assessment: All subjects will rate their average pain intensity using a VAS pain scale. The assessment will perform before the first use of PCA or supplemental analgesics and at 4±1, 24±2, 32±3, 48±4 hours and once daily on Days 3 to Day 5 after the surgery.
* Brief Pain Inventory (BPI) will be evaluated at Day 2.
* Vital signs (temperature, respiratory rate, blood pressure and heart rate) will be checked once daily before Day 6.
* In Group 1 (NALDEBAIN group), the injection site will be evaluated once daily before final visit.
* Review of concomitant medication and adverse event record.
* In Group 2 (PCA group), the amount of fentanyl used will be recorded on Days 0 through 2.

Study Day 6 Evaluate the following items at Day 6.

* Pain assessment: Subjects will rate their pain intensity in the patient diary.
* Brief Pain Inventory (BPI) will be evaluated.
* Vital signs (temperature, respiratory rate, blood pressure and heart rate) will be checked.
* Injection site evaluation.
* Review of the adverse event record.
* Review of concomitant medication. Final Visit (Day of Discharge, Day 6~30)
* Vital signs (temperature, respiratory rate, blood pressure and heart rate) will be checked
* Injection site evaluation
* Laboratory tests, including hematological and biochemical tests, and urinalysis.
* Patient satisfaction: At the final visit, each subject was asked the following question: "How satisfied were you with your postsurgical analgesia"? Subjects were asked to classify themselves as either "highly satisfied", "satisfied", "uncertain", "dissatisfied", or "very dissatisfied".
* Physical examination.
* Review of the adverse event record.
* Review of concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is among 20 to 80 years of age at screening.
* Scheduled to electively undergo open-laparotomy.
* American Society of Anesthesiology Physical Class 1-3.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Body mass index less than 18 kg/m2 or greater than 30 kg/m2.
* History of previous open-laparotomy.
* Surgery with major complication, or need blood transfusion.
* History of hypersensitivity or adverse reaction to local anesthetics, opioid, or any ingredient of the medications administered in this study.
* Severe comorbidity.
* Chronic preoperative opioid consumption.
* Pregnant or breastfeeding.
* Inability to use the PCA device.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
pain assessment (post-OP 48 hours) | During post-OP 48 hours
  Pain assessment (time-specific pain intensity) calculated as the area under the curve of VAS pain intensity scores through 48 hours after surgery.

SECONDARY OUTCOMES:
supplemental analgesics | From post-OP to Day 6
  The consumption of total amount (mg) of supplemental analgesics administered after surgery.
Pain assessment (post-OP to Day 6) | From post-OP to Day 6
  Pain assessment calculated as the area under the curve of VAS pain intensity scores through end of surgery to Day 6
Brief Pain Inventory | pre-OP Day -1, post-OP Day 2 and Day 6
  Pain intensity and interference of Brief Pain Inventory (BPI)
Patient satisfaction | On discharge Day, between post-OP Day 7 and Day 14
  Patient satisfaction on a 5-point rating.
Length of postoperative hospital stay | From post-OP to Discharge Day, about 1 to 2 weeks
  Length of postoperative hospital stay.

OTHER OUTCOMES:
Adverse event | From post-OP Day 1 to Discharge Day, about 1 to 2 weeks
  Incidence of treatment-emergent adverse event (TEAE)
other abnormalities | From Screening Day to Discharge Day, about 1 to 2 weeks
  Percentage of abnormal from baseline to final visit in vital signs, laboratory tests and injection site evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, PhD, Study Chair — Division of Colorectal Surgery, Department of Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang TK, Huang CW, Su WC, Tsai HL, Ma CJ, Yeh YS, Chen YC, Li CC, Cheng KI, Su MP, Wang JY. Extended-Release Dinalbuphine Sebacate Versus Intravenous Patient-Controlled Analgesia with Fentanyl for Postoperative Moderate-to-Severe Pain: A Randomized Controlled Trial. Pain Ther. 2020 Dec;9(2):671-681. doi: 10.1007/s40122-020-00197-x. Epub 2020 Sep 29. PMID 32990938
- [Derived] Tsai HL, Chang TK, Su WC, Yeh YS, Huang CW, Ma CJ, Wang JY. Comparing efficacy and safety between Naldebain(R) and intravenous patient-controlled analgesia with fentanyl for pain management post-laparotomy: study protocol for a randomized controlled, non-inferior trial. Trials. 2019 Mar 18;20(1):173. doi: 10.1186/s13063-019-3260-4. PMID 30885242